CLINICAL TRIAL: NCT03081104
Title: Comparative Study Between Operative Hysteroscopy Versus the Ultrasound Guided Vacuum Aspiration Versus the Blind Vacuum Aspiration for the Treatment of the Missed Abortion
Brief Title: Operative Hysteroscopy and Ultrasound Guided Vacuum Aspiration Versus Blind Vacuum Aspiration for the Treatment of Missed Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hystroscopy (Active Comparator): The procedure will be performed by a gynecological surgeon, under general anaesthesia with the patient in lithotomy position. Antibiotic prophylaxis may be administered, the cervix is grasped with pozzi forceps and dilated up to hegar 9 to facilitate insertion of the hysteroscopy. The uterine cavity will be distended with saline or glycine, depending on the polarity of the resection system.with a maximum irrigation pressure of 110mmHg. The retained products will be resected from top to bottom with surgical resector without electric power. The use of forceps or curettes to facilitate the removal of material is permitted. If active bleeding occurs , elective coagulation by hystroscope is done to stop intrauterine bleeding. The deficit of distending media should be calculated at the end of procedure.
  Interventions: Device: hystroscopy
- ultrasound guided aspiration (Active Comparator): The transducer was held on the abdomen to obtain a longitudinal image of the uterus and cervix and provide the surgeon with a visual reference of the gestational sac, cervical canal and any instruments passed into the uterus.The progress of the operation was continuously monitored as the uterine contents were evacuated under visual control. It was possible to keep the dilators and the suction cannula under constant view by slightly tilting the transducer as required. Advancement of any instrument was allowed only under direct ultrasound control.The completeness of the evacuation was confirmed by the scan in these cases.
  Interventions: Device: ultrasound; Procedure: Aspiration
- blind aspiration (Active Comparator): The women were allowed to empty their urinary bladder before induction of anesthesia, but catheterization was not performed. After positioning the patient appropriately on the operating table, bimanual pelvic examination was performed under anesthesia to assess the axis and the size of the uterus. A Sim's speculum was inserted into the vagina; the cervix was visualized and grasped using the Vulsellum forceps. The cervical canal was dilated gradually with Hegar dilators up to the size corresponding to the weeks of gestation. The uterine cavity was evacuated using a plastic cannula attached to an electric suction apparatus. Negative pressure of 75 mmHg was used. The aspirate was examined to confirm the presence of products of conception. The completeness of the evacuation was checked by gentle sharp curettage and final suctioning at the end of procedure.
  Interventions: Procedure: Aspiration

INTERVENTIONS:
Device: hystroscopy — The uterine cavity will be distended with saline or glycine, depending on the polarity of the resection system.with a maximum irrigation pressure of 110mmHg. The retained products will be resected from top to bottom with surgical resector without electric power. The use of forceps or curettes to facilitate the removal of material is permitted. If active bleeding occurs , elective coagulation by hystroscope is done to stop intrauterine bleeding. The deficit of distending media should be calculated at the end of procedure.
  Arms: hystroscopy
Device: ultrasound — The transducer was held on the abdomen to obtain a longitudinal image of the uterus and cervix and provide the surgeon with a visual reference of the gestational sac, cervical canal and any instruments passed into the uterus.The progress of the operation was continuously monitored as the uterine contents were evacuated under visual control.
  Arms: ultrasound guided aspiration
Procedure: Aspiration — The cervical canal was dilated gradually with Hegar dilators up to the size corresponding to the weeks of gestation. The uterine cavity was evacuated using a plastic cannula attached to an electric suction apparatus. Negative pressure of 75 mmHg was used.
  Arms: blind aspiration; ultrasound guided aspiration

SUMMARY:
The intervention to be evaluated are operative hysteroscopy(group A) and ultrasound guided aspiration(group C) and blinded vacuum aspiration(group B).

For all surgical procedures , surgical antibiotics prophylaxis, misoprostol to dilate cervix, and anti adhesion barrier gel will be used. The evacuated retention products will be sent for pathological examination.

Group A: Operative Hystroscopy:

The procedure will be performed under general anaesthesia with the patient in lithotomy position. the cervix is grasped with pozzi forceps and dilated up to hegar 9 to facilitate insertion of the hysteroscopy. The uterine cavity will be distended with saline or glycine, with a maximum irrigation pressure of 110mmHg. The retained products will be resected from top to bottom with surgical resector without electric power. The use of forceps or curettes to facilitate the removal of material is permitted. .

Group B:blinded vacuum aspiration of gestational contents:

The women were allowed to empty their urinary bladder before induction of anesthesia, After positioning the patient appropriately on the operating table, bimanual pelvic examination was performed under anesthesia to assess the axis and the size of the uterus. A Sim's speculum was inserted into the vagina; the cervix was visualized and grasped using the Vulsellum forceps. The cervical canal was dilated gradually with Hegar dilators up to the size corresponding to the weeks of gestation. The uterine cavity was evacuated using a plastic cannula attached to an electric suction apparatus. Negative pressure of 75 mmHg was used. The aspirate was examined to confirm the presence of products of conception. The completeness of the evacuation was checked by gentle sharp curettage and final suctioning at the end of procedure.

Group C: Ultrasound guided aspiration curettage :

same as group B but guided with ultrasound

DETAILED DESCRIPTION:
The intervention to be evaluated are operative hysteroscopy(group A) and ultrasound guided aspiration(group C) and blinded vacuum aspiration(group B).these procedures are routinely performed in the obstetrics and gynecology department for various indications. For all surgical procedures , surgical antibiotics prophylaxis, misoprostol to dilate cervix, and anti adhesion barrier gel will be used. The evacuated retention products will be sent for pathological examination. RH negative women will receive prophylaxis to prevent RH alloimmunization.

Group A: Operative Hystroscopy:

The procedure will be performed by a gynecological surgeon, under general anaesthesia with the patient in lithotomy position. Antibiotic prophylaxis may be administered, the cervix is grasped with pozzi forceps and dilated up to hegar 9 to facilitate insertion of the hysteroscopy. The uterine cavity will be distended with saline or glycine, depending on the polarity of the resection system.with a maximum irrigation pressure of 110mmHg. The retained products will be resected from top to bottom with surgical resector without electric power. The use of forceps or curettes to facilitate the removal of material is permitted. If active bleeding occurs , elective coagulation by hystroscope is done to stop intrauterine bleeding. The deficit of distending media should be calculated at the end of procedure.

Group B:blinded vacuum aspiration of gestational contents:

The women were allowed to empty their urinary bladder before induction of anesthesia, but catheterization was not performed. After positioning the patient appropriately on the operating table, bimanual pelvic examination was performed under anesthesia to assess the axis and the size of the uterus. A Sim's speculum was inserted into the vagina; the cervix was visualized and grasped using the Vulsellum forceps. The cervical canal was dilated gradually with Hegar dilators up to the size corresponding to the weeks of gestation. The uterine cavity was evacuated using a plastic cannula attached to an electric suction apparatus. Negative pressure of 75 mmHg was used. The aspirate was examined to confirm the presence of products of conception. The completeness of the evacuation was checked by gentle sharp curettage and final suctioning at the end of procedure.

Group C: Ultrasound guided aspiration curettage :

The transducer was held on the abdomen to obtain a longitudinal image of the uterus and cervix and provide the surgeon with a visual reference of the gestational sac, cervical canal and any instruments passed into the uterus.The progress of the operation was continuously monitored as the uterine contents were evacuated under visual control. It was possible to keep the dilators and the suction cannula under constant view by slightly tilting the transducer as required. Advancement of any instrument was allowed only under direct ultrasound control.The completeness of the evacuation was confirmed by the scan in these cases.

ELIGIBILITY:
Inclusion Criteria:

- Women in the fertility perioddiagnosed with missed abortion in the first trimester < 14 wks of gestation.

The pregnancy concerned should correspond to a planned or wanted baby. Diagnosis of missed abortion by transvaginal ultrasound showing sgestational sac with no cardiac pulsations.

Exclusion Criteria:

* • Other type of abortion.

  * Known uterine malformation.
  * History of surgical intervention done in the uterus or uterine cavity.
  * Moderate to sever vaginal bleeding needing rapid surgical intervention.
  * Presence of IUD
  * Current pregnancy obtained by IVF cycle
  * Extrauterine pregnancy

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate after evacuation | 12 months after procedure
  duration needed to achieve pregnancy after evacuation provided non use of contraceptive methods

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Meshaal H, Salah E, Fawzy E, Abdel-Rasheed M, Maged A, Saad H. Hysteroscopic management versus ultrasound-guided evacuation for women with first-trimester pregnancy loss, a randomised controlled trial. BMC Womens Health. 2022 May 25;22(1):190. doi: 10.1186/s12905-022-01774-2. PMID 35614405